CLINICAL TRIAL: NCT06815003
Title: Phase-2 Study of Vedolizumab Plus Post-Transplant Cyclophosphamide and Short Course Tacrolimus for Graft-versus-Host Disease Prevention After Reduced Intensity Conditioning Peripheral Blood Stem Cell Allogeneic Hematopoietic Cell Transplantation
Brief Title: Vedolizumab Plus Post-transplant Cyclophosphamide and Short Course Tacrolimus for the Prevention of Graft Versus Host Disease in Patients Undergoing Allogeneic Hematopoietic Cell Transplantation After Reduced Intensity Conditioning
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24473; NCI-2025-00341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24473 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-02-07 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Graft Versus Host Disease; Myelodysplastic Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Graft vs Host Disease; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Stem Cell Transplantation; Specimen Handling; Biopsy; Cyclophosphamide; fludarabine; Melphalan; Tacrolimus; vedolizumab; Immunoglobulin G; Disulfides; LDP-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (vedolizumab, cyclophosphamide, tacrolimus) (Experimental): Patients receive reduced intensity conditioning with fludarabine IV on days -7 to -3 and melphalan IV on day -2. Patients then undergo allogeneic HCT on day 0. Patients also receive vedolizumab IV over 30 minutes on days -1, +13, +41, +69, +97, +125, and +153, cyclophosphamide IV on days +3 and +4, and tacrolimus IV or PO on day +5 to day +95 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT and ECHO or MUGA during screening, blood sample collection on study, and bone marrow biopsy throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Tacrolimus; Biological: Vedolizumab

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Questionnaire Administration — Ancillary studies
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Biological: Vedolizumab — Given IV
  Other Names: Entyvio; Immunoglobulin G1, anti-(human integrin LPAM-1 (lymphocyte Peyer's patch adhesion molecule 1)) (human-Mus musculus heavy chain), disulfide with human-Mus musculus kappa-chain, dimer; LDP 02; LDP-02; LDP02; MLN0002; MLN02

SUMMARY:
This phase II trial studies how well vedolizumab plus post-transplant cyclophosphamide (PTCy) and short course tacrolimus work for the prevention of graft versus host disease (GVHD) in patients undergoing allogeneic hematopoietic cell transplantation (HCT) after reduced intensity conditioning. Allogeneic HCT is a procedure in which a person receives blood-forming stem cells (cells from which all blood cells develop) from a donor. Giving reduced conditioning chemotherapy before an allogeneic HCT helps kill cancer cells in the body and helps make room in the patient's bone marrow for new stem cells to grow using less than standard doses of chemotherapy. Sometimes, the transplanted cells from a donor can attack the body's normal cells (called graft-versus-host disease). Vedolizumab is a monoclonal antibody, which is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). It may reduce inflammation. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid and may kill cancer cells. It may also lower the body's immune response. Tacrolimus suppresses the immune system by preventing the activation of certain types of immune cells. Giving vedolizumab plus PTCy and short course tacrolimus may be effective at preventing GVHD after allogeneic HCT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and describe the toxicity profile of adding vedolizumab at a fixed dose level to post-transplant cyclophosphamide (PTCy) -based graft-versus-host disease (GVHD) prophylaxis with tacrolimus after mobilized peripheral blood stem cell (PBSC) allogeneic hematopoietic cell transplantation (HCT) from a matched related/unrelated donor. (Safety lead-in segment) II. Assess the efficacy of vedolizumab in combination with PTCy by grade 2-4 acute GVHD-free survival by day+180 after allogeneic hematopoietic cell transplantation (HCT). (Expansion segment)

SECONDARY OBJECTIVES:

I. Continue safety assessment of vedolizumab + PTCy combination as GVHD prophylaxis in the expansion cohort.

II. Estimate overall survival (OS), progression-free survival (PFS), cumulative incidences of relapse/disease progression, and non-relapse mortality (NRM) at 100 days, and 1-year post-transplant.

III. Estimate rates of acute GVHD (day 100 and 180 post-HCT), lower gastrointestinal (GI) GVHD (day 100 and day 180 post-HCT), chronic GvHD (1-year post-HCT), infections (100 and 180 days and 1 year post HCT).

IV. Estimate rates of complete remission, and neutrophil recovery. V. Evaluate and describe the cytokine release syndrome (CRS) post-HCT by assessing the incidence, frequency, and severity of CRS.

EXPLORATORY OBJECTIVES:

I. Donor cell engraftment will be assessed by count monitoring and short tandem repeat (STR) chimerism analysis on days +30 and day +100.

II. Describe the kinetics of immune cell recovery. III. Evaluate patient's quality of life on day +100, 6 months and one-year post-HCT.

IV. Describe the kinetics of GVHD biomarkers, and inflammatory cytokines for up to 100 days post-HCT.

V. Obtain a preliminary estimate of gut microbiome diversity at baseline (preferably before fludarabine administration), and then on days +14, +30, +60, +100, and +180 after HCT.

OUTLINE:

Patients receive reduced intensity conditioning with fludarabine intravenously (IV) on days -7 to -3 and melphalan IV on day -2. Patients then undergo allogeneic HCT on day 0. Patients also receive vedolizumab IV over 30 minutes on days -1, +13, +41, +69, +97, +125, and +153, cyclophosphamide IV on days +3 and +4, and tacrolimus IV or orally (PO) on day +5 to day +95 in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) and echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening, blood sample collection on study, and bone marrow biopsy throughout the study.

After completion of study treatment, patients are followed up at 30 days after the last dose of vedolizumab, day +180 and at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 and ≤ 80 years old

  * Note: Patients > 70 years of age must have Karnofsky performance status ≥ 80 and hematopoietic cell transplantation-comorbidity index (HCT-CI) ≤ 2
* Karnofsky performance status ≥ 70%
* Patients with the following diagnosis, eligible to undergo allogeneic HCT from an 8/8 match related/unrelated donor (A, B, C, DR by high resolution typing)

  * Acute Leukemias (acute myeloid leukemia [AML] or acute lymphoblastic leukemia [ALL]) in complete remission with bone marrow (BM) blast of < 5%
  * Myelodysplastic syndrome (blast < 10%)
  * Myeloproliferative neoplasm (MPN) other than myelofibrosis (MF) needing HCT
  * Chronic myelomonocytic leukemia (CMML)
* Hemoglobin ≥ 9g/dL (within 30 days prior to day 1 of protocol therapy)

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 2.0 mg/dL (unless has Gilbert's disease) AND serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) < 5 times the upper limit of normal (ULN) (within 30 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 3.0 x ULN (within 30 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 3.0 x ULN (within 30 days prior to day 1 of protocol therapy)
* Creatinine clearance of ≤ 1.5 mg/dL or ≥ 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 30 days prior to day 1 of protocol therapy)
* Left ventricular ejection fraction (LVEF) ≥ 50%

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* IF ABLE TO PERFORM PULMONARY FUNCTION TESTS: Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and DLCO (diffusion capacity) ≥ 50% of predicted (corrected for hemoglobin)

  * Note To be performed within 28 days prior to day 1 of protocol therapy
* IF UNABLE TO PERFORM PULMONARY FUNCTION TESTS: Oxygen (O2) saturation > 92% on room air

  * Note To be performed within 28 days prior to day 1 of protocol therapy
* Seronegative for HIV antigen/antibody (Ag/Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative) (within 30 days prior to day 1 of protocol therapy)

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Tuberculosis test (within 30 days prior to day 1 of protocol therapy)

  * Patients with positive tuberculosis (TB) test results will have infectious disease (ID) evaluation and post HCT therapy with isoniazid (INH) for 6 months with ID follow up. Vaccinated patients will need negative chest X-ray results
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test (within 30 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior allogeneic HCT
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 14 days prior to day 1 of protocol therapy

  * Note: Conditioning regimen within 14 days prior to day 1 of protocol therapy is not considered as an exclusion criterion. Patients on maintenance chemotherapy with agents listed are not excluded
* Other investigational drugs for GVHD prophylaxis
* Herbal medications
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Active infection not responding to antibiotics
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Females only: Pregnant or breastfeeding
* Patients not expected to be available for follow-up in our institution for at least 100 days after the transplant
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary engraftment failure (Safety lead-in segment) | From starting the first dose of vedolizumab to the first observation of event, day +30, whichever comes first
  Will be assessed as an unacceptable toxicity (UT). Will include type, severity, duration, and attribution/association with the study regimen and dose limiting toxicity (DLT) occurrence. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including, but not limiting infections, other adverse events of special interest, and severe adverse events. Point estimates and corresponding exact 90% confidence intervals (CIs) will be provided for each measure of toxicity/adverse events.
Incidence of severe infusion reaction (Safety lead-in segment) | From starting the first dose of vedolizumab to the first observation of event, day +30, whichever comes first
  Will be assessed as a UT. Will assess severe infusion reactions, grade 4 per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0, after receiving the 1st or 2nd dose of vedolizumab. Will include type, severity, duration, and attribution/association with the study regimen and DLT occurrence. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including, but not limiting infections, other adverse events of special interest, and severe adverse events. Point estimates and corresponding exact 90% CIs will be provided for each measure of toxicity/adverse events.
Incidence of grade 4-5 adverse events (Safety lead-in segment) | From starting the first dose of vedolizumab to the first observation of event, day +30, whichever comes first
  Will be assessed as a UT. Will assess grade 4-5 adverse events based on CTCAE v 5.0 probably or definitely attributable to vedolizumab. Will include type, severity, duration, and attribution/association with the study regimen and DLT occurrence. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including, but not limiting infections, other adverse events of special interest, and severe adverse events. Point estimates and corresponding exact 90% CIs will be provided for each measure of toxicity/adverse events.
Non-relapse mortality (NRM) (Safety lead-in segment) | From date of stem cell infusion until non-disease related death, assessed up to 1 year post-hematopoietic cell transplant (HCT)
  Will be assessed as a UT. Defined as death occurring in a patient from causes other than relapse or progression. Deaths from relapse/progression will be considered a competing risk. NRM will be censored at last follow-up if patients are alive and remain disease free. Will be analyzed using the Kaplan-Meier curves.
Incidence of grade 2-4 acute graft versus host disease (GVHD)-free survival | From start of HCT to first occurrence of grade 2-4 acute GVHD followed until day +180 or death from any cause, whichever occurs first, assessed up to 1 year post-HCT
  Will be assessed among patients in the safety lead-in and dose expansion segments. Will be estimated using Kaplan-Meier curve.

SECONDARY OUTCOMES:
Incidence of adverse events (Expansion segment) | From the start of first dose of vedolizumab to day +130 post-HCT
  Will be assessed using CTCAE v5.0. Will assess grade 4-5 adverse events probably or definitely attributable to study regiment by day +30 post-HCT and grade 3-5 adverse events probably or definitely attributed to study regimen by day +130 that are not UT. Will include type, severity, duration, and attribution/association with the study regimen and DLT occurrence. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including, but not limiting infections, other adverse events of special interest, and severe adverse events. Point estimates and corresponding exact 90% CIs will be provided for each measure of toxicity/adverse events.
Incidence of grade 3-5 adverse events at least probably attributable to vedolizumab, but not UT | Up to day +180 post-HCT
  Will be assessed using CTCAE v5.0. Will include type, severity, duration, and attribution/association with the study regimen and DLT occurrence. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including, but not limiting infections, other adverse events of special interest, and severe adverse events. Point estimates and corresponding exact 90% CIs will be provided for each measure of toxicity/adverse events.
Overall survival | From the day of stem cell infusion until death, assessed up to 1 year post-HCT
  Patients are considered a failure for this endpoint if they die, regardless of cause. Will be censored at last follow-up if the last known status is alive. Will be analyzed using the Kaplan-Meier curves.
Progression free survival | From the date of stem cell infusion to the date of death, disease relapse/progression, whichever occurs first, assessed up to 1 year post-HCT
  Patients are considered a failure for this endpoint if they die (regardless of cause) or experience disease progression or relapse. Will be censored at last follow-up if patients are alive and remain disease free. Will be analyzed using the Kaplan-Meier curves.
Relapse/progression rate | From day of stem cell infusion (day 0) to 1 year post-HCT
  Deaths without relapse/progression will be considered a competing risk. Surviving patients with no history of relapse/progression will be censored at time of last follow-up. Will be analyzed using the Kaplan-Meier curves.
NRM | From date of stem cell infusion until non-disease related death, assessed up to 1 year post-HCT
  Defined as death occurring in a patient from causes other than relapse or progression. Deaths from relapse/progression will be considered a competing risk. NRM will be censored at last follow-up if patients are alive and remain disease free. Will be analyzed using the Kaplan-Meier curves.
Incidence of acute GVHD | From day 0 to days +100 and +180 post-HCT
  Will be graded and staged according to Mount Sinai Acute GVHD International Consortium (MAGIC) criteria. The first day of acute GVHD onset at a certain grade will be used to calculate the cumulative incidence (grades II-IV). Will be evaluated among all patients treated with study regimen. Will be estimated using Kaplan-Meier curve.
Incidence of lower gastrointestinal GVHD | From day 0 to days +100 and +180 post-HCT
  Will be graded and staged according to MAGIC criteria. The first day of acute GVHD onset at a certain grade will be used to calculate the cumulative incidence (grades II-IV). Will be evaluated among all patients treated with study regimen. Will be estimated using Kaplan-Meier curve.
Incidence chronic GVHD | From day +80 post-HCT to 1 year post-HCT
  Will be evaluated and scored according to National Institutes of Health Consensus Staging. The first day of chronic GVHD onset will be used to calculate the cumulative incidence. Will be evaluated among all patients treated with study regimen. Will be estimated using Kaplan-Meier curve.
Incidence of infections | At days +100 and +180 post-HCT and 1 year post-HCT
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.
Hematologic recovery | Up to 1 year post-HCT
  Will be defined as absolute neutrophil count (ANC) ≥ 0.5 x 10^3/μL achieved and sustained for 3 consecutive lab values on different days with no subsequent decline and platelets ≥ 20 K/μL independent of platelet transfusion support (date should reflect no transfusions in previous 7 days, and the first of 3 consecutive lab values on different days).
Primary graft failure | Up to 28 days post-HCT
  Will be defined as failure to achieve ANC of 500 or more for 3 days and, hypocellular marrow, and donor chimerism of < 5% all by day 28.
Incidence of cytokine release syndrome | Up to 1 year post-HCT
  Will be defined and graded per American Society for Transplantation and Cellular Therapy criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M. Al Malki, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States